CLINICAL TRIAL: NCT03708406
Title: Otologic and Rhinologic Outcomes in Children With Cleft Palate at Age 10 Years
Brief Title: Otologic and Rhinologic Outcomes in Children With Clef Palate
Acronym: Clef Palate
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0374
Record Dates: First submitted 2018-10-08; First posted 2018-10-17 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cleft Lip and Palate
Keywords: cleft palate; Eustachian dysfunction; Obstructive ventilation
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Middle ear effusion fluids
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Cleft lip and palate: Children with Cleft lip and palate
- Children with Cleft palate: Children with Cleft palate

SUMMARY:
OBJECTIVE:

To compare otologic and rhinologic outcomes in patients with cleft palate according to surgical protocols and type of cleft.

DESIGN:

Monocentric retrospective and prospective analysis of medical reports.

PATIENTS, PARTICIPANTS:

All consecutively treated patients affected by a cleft palate, born between December 2006 and December 2009 and followed in the Montpellier University Hospital, at the age of 10 years.

INTERVENTIONS:

Results of audiometry, tympanometry, otoscopy, tubomanometry and rhinomanometry and orofacial tomodensitometry done at the age of 10 were evaluated.

MAIN OUTCOME MEASURE(S):

The history of ventilation tubes inserted, and the results at the EDTQ test were analyzed.

ELIGIBILITY:
Inclusion criteria :

* 10 yo children with operated clefts followed in the universitary hospital of Montpellier
* who went to the ENT check up

Exclusion criteria :

* Thoses who skip the check up

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutively treated patients affected by a cleft lip and palate or a cleft palate, born between December 2006 and December 2009 and followed in the Montpellier University Hospital, at the age of 10 years.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Audiometry | 1 day
  evaluation of the hearing threshold

SECONDARY OUTCOMES:
nasal ventilation | 1 day
  Nasal ventilation will be assessed with passive anterior rhinomanometry
Eustachian tube function | 1 day
  Eustachian tube function will be assessed with tubomanometry
Facial 3D scan | 1 day
  Facial 3D scan will be used to measure 2 criteria :
  * Total volum of the mastoid
  * Total volum of the mastoid's cells (pneumatization)
  Facial 3D scan will be used to measure 2 criteria :
  * Total volum of the mastoid
  * Total volum of the mastoid's cells (pneumatization)
  Facial 3D scan will be used to measure 2 criteria :
  * Total volum of the mastoid
  * Total volum of the mastoid's cells (pneumatization)

CONTACTS AND LOCATIONS:
Overall Officials: Lylou Casteil Baume, ENT resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France